CLINICAL TRIAL: NCT03311659
Title: Evaluation of Immunogenicity, Safety and Reactogenicity of GSK Biologicals' dTpa Booster Vaccine (263855) (Boostrix) Administered as a Booster Dose in Healthy Russian Subjects
Brief Title: Evaluation of Immunogenicity, Safety and Reactogenicity of GSK Biologicals' Boostrix Vaccine Administered as a Booster Dose in Healthy Russian Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201532; 2015-003405-42 (EudraCT Number)
Record Dates: First submitted 2017-10-06; First posted 2017-10-17 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Diphtheria-Tetanus-acellular Pertussis Vaccines
Keywords: Diphtheria; Pertussis; Tetanus; Immunogenicity
MeSH Terms: conditions — Diphtheria; Whooping Cough; Tetanus | interventions — Boostrix

STUDY DESIGN:
Masking Description: The treatment allocation would be non-randomised and stratified by age into four strata [4-9 years (children), 10-17 years (adolescents), 18-64 (adults) years and ≥65 years (elderly population)].
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dTpa group (Experimental): Healthy female and male subjects with age 4 years and above and who received a single dose of Boostrix vaccine at Day 1.
  Interventions: Biological: Boostrix

INTERVENTIONS:
Biological: Boostrix — One dose administered intramuscularly in the deltoid muscle of the non-dominant arm in dTap group.

SUMMARY:
Diphtheria, tetanus and pertussis are common causes of diseases worldwide, with significant morbidity and mortality. The purpose of this study is to assess the immunogenicity, safety and reactogenicity of a single dose of GlaxoSmithKline (GSK) Biologicals' Boostrix vaccine, administered as a booster dose in healthy Russian subjects. An equal number of subjects are expected to be recruited in the following age categories: 4-9 years (children), 10-17 years (adolescents), 18-64 years (adults) and ≥65 years (elderly population). By receiving the Boostrix vaccine, the subjects could be protected against diphtheria, tetanus and pertussis diseases.

DETAILED DESCRIPTION:
The study is a phase III, open-label, self-contained, multi-centre, uncontrolled, single-country study with a single group. Treatment will be allocated in a non-randomised process and stratified by age as 4-9 years (children), 10-17 years (adolescents), 18-64 years (adults) and ≥65 years (elderly population). The study will consist of a single primary epoch (001) starting at Visit 1 (Day 1) with the administration of a single dose of Boostrix vaccine and ending at Visit 2 (Day 31). Blood samples will be collected at Visits 1 and 2.

Protocol Amendment 1 was developed to implement the following changes:

* Wording "parents/Legally Acceptable Representative(s) (LAR[s])" was replaced by the wording "parent(s)/adoptive parent(s)". As per Russian legislation, only parents or adoptive parents can give consent for the enrolment of their child in a clinical trial. No other person is allowed to give consent on behalf of a minor to participate in a clinical trial.
* The age groups at inclusion to study were amended according to the approved Boostrix EU label and physiological particularities i.e., from 3-9 to 4-9 years (children), 10-19 to 10-17 years (adolescents), 20-64 to 18-64 years (adults) and ≥65 years (elderly population).
* The inclusion criteria have been amended in order to clarify the following,

  * Children from four to seven years of age who have received diphtheria, tetanus and pertussis vaccination prior to study enrolment as per local recommendations will be enrolled
  * Subjects eight years of age and older who have received diphtheria, tetanus and pertussis vaccination to the best of their/subjects' parent(s)/subjects' adoptive parent(s) knowledge and did not receive an additional diphtheria, tetanus or pertussis vaccination within five years prior to enrolment in the study will be enrolled.

Protocol amendment 2 was developed after the comments from the Russian regulatory authorities [Ministry of Health (MoH)]. Adjustments to the text were made to clarify the inclusion and exclusion criteria for enrolment of subjects and the conduct of the study. In addition, adjustments for the reporting period and assessment of adverse events in the safety sections were made for consistency. The newly re-developed and re-validated GSK's DTPa ELISA cut-offs were updated as per the most recent CBER recommendation (2017).

Protocol amendment 3 is developed to accommodate older adults (approximately 58 years old and older) who were born before national recommendations in Russia for infant DTP vaccination. Adjustments to the text are made in the inclusion criteria to clarify the enrolment of subjects for age group eight years and above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or subjects' parent(s)/adoptive parent(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female four years of age and older.
* Written informed consent obtained from the subject/from the parent(s)/adoptive parent(s) of the subject prior to performing any study specific procedure.
* Written informed assent obtained from subjects aged 14 years to <18 years.
* Healthy subjects as established by medical history and physical examination before entering into the study.
* Children 4-7 years of age with documented previous diphtheria, tetanus and pertussis vaccination (primary series and first booster) as per local recommendation prior to study enrolment, but should have not received any further diphtheria-tetanus containing booster planned at 6-7 years of age as per local recommendations or any other diphtheria, tetanus and pertussis containing vaccine.
* Subjects eight years of age and older who can report previous diphtheria, tetanus with or without pertussis vaccination - documented or to the best of their/subjects' parent(s)/subjects' adoptive parent(s) knowledge - and did not receive an additional diphtheria, tetanus with or without pertussis vaccination within five years prior to enrolment in the study will be enrolled.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception within 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the vaccination.

Exclusion Criteria:

* Child in care
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* History of previous or intercurrent diphtheria, tetanus or pertussis diseases since birth in subjects four to seven years of age.
* History of previous or intercurrent diphtheria, tetanus or pertussis diseases within 5 years prior to enrolment in subjects aged eight years and above.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day (for adult subjects, ≥18 years of age) or ≥ 0.5 mg/kg/day (for paediatric subjects, aged 4-17 years), or equivalent. Inhaled and topical steroids are allowed
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after the dose of vaccine with the exception of inactivated influenza vaccine which can be given at any time during the study conduct as per the Summary of Product Characteristics (SPC) and according to the local governmental recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* History of encephalopathy after administration of a previous dose of pertussis vaccine that could not be attributed to another identifiable cause, progressive neurologic disorder, uncontrolled epilepsy or progressive encephalopathy: pertussis vaccine should not be administered to individuals with these conditions until a treatment regimen has been established and the condition has stabilised.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥38.0°C. The preferred location for measuring temperature in this study will be the axilla.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant uncontrolled pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination and/or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions during the study conduct.
* Any medical condition that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Russia (7):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Murmansk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20721

REFERENCES:
- [Background] Asatryan A, Meyer N, Scherbakov M, Romanenko V, Osipova I, Galustyan A, Shamsheva O, Latysheva T, Myasnikova T, Baudson N, Dodet M, Xavier S, Harrington L, Kuznetsova A, Campora L, Van den Steen P. Immunogenicity, safety, and reactogenicity of combined reduced-antigen-content diphtheria-tetanus-acellular pertussis vaccine administered as a booster vaccine dose in healthy Russian participants: a phase III, open-label study. Hum Vaccin Immunother. 2021 Mar 4;17(3):723-730. doi: 10.1080/21645515.2020.1796423. Epub 2020 Aug 26. PMID 32845735

RESULTS

PARTICIPANT FLOW:
Groups:
- dTpa Group: Healthy female and male subjects aged 4 years and above, who received a single dose of Boostrix vaccine at Day 1.
Period: Overall Study
Arm/Group | dTpa Group
Started | 447
Completed | 446
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | dTpa Group
Number analyzed (Participants) | 447
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (27.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241
  Male | 206
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian / European Heritage | 447

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects for Anti-diphtheria (Anti-D).
Description: A seroprotected subject was a subject whose anti-D concentrations were greater than or equal to (≥) 0.1 International units per milliliter (IU/ml). Seroprotection was assessed by enzyme-linked immunosorbent assay (ELISA) method. In addition, sera with ELISA concentrations <0.1 IU/ml were tested for neutralising antibodies using a Vero-cell neutralisation assay. Both the ELISA test (antibody concentrations ≥ 0.1 IU/ml) and Vero-cell test (antibody concentration ≥ 0.01 IU/ml) defined the seroprotection status for the primary endpoint.
Time Frame: At Day 31
Population: The Per Protocol (PP) Cohort for immunogenicity included all evaluable subjects who had received the dose of study vaccine, met all eligibility criteria, complied with the procedures and intervals defined in the protocol, for whom assay results were available for antibodies against at least one study vaccine antigen component.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 441
Participants
  Anti-D antibody ≥ 0.1 IU/ml: number analyzed (Participants) | 438
  Anti-D antibody ≥ 0.1 IU/ml | 437
  Neutralizing anti-D antibody ≥ 0.01 IU/ml: number analyzed (Participants) | 1
  Neutralizing anti-D antibody ≥ 0.01 IU/ml | 1

2. Primary Outcome: Number of Seroprotected Subjects for Anti-tetanus (Anti-T).
Description: A seroprotected subject was a subject whose anti-T concentrations were ≥ 0.1 IU/ml. Seroprotection was assessed by ELISA method.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 441
Participants | 439

3. Primary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN).
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal to the assay cut-off value. Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN respectively.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 442
Participants
  Anti-PT antibody: number analyzed (Participants) | 440
  Anti-PT antibody | 430
  Anti-FHA antibody | 442
  Anti-PRN antibody: number analyzed (Participants) | 436
  Anti-PRN antibody | 431

4. Secondary Outcome: Number of Subjects With a Booster Response to the Diphtheria and Tetanus Antigens
Description: Booster response to diphtheria (D) and tetanus (T) antigens was defined according to pre-vaccination antibody concentration:
  1. for subjects with values <0.1 IU/ml (i.e. below the seroprotection cut-off), antibody concentrations of at least ≥0.4 IU/ml, one month after vaccination; and
  2. for subjects with values ≥0.1 IU/ml (i.e. equal to or above the seroprotection cut-off), an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination. Seronegative (S-) subjects are those who have antibody concentration less than (<) 0.1 IU/mL and seropositive (S+) subjects are those who have antibody concentration ≥ 0.1 IU/mL prior to vaccination.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 441
Participants
  Anti-D antibody, S-: number analyzed (Participants) | 33
  Anti-D antibody, S- | 26
  Anti-D antibody, S+: number analyzed (Participants) | 398
  Anti-D antibody, S+ | 282
  Anti-D antibody, Overall: number analyzed (Participants) | 431
  Anti-D antibody, Overall | 308
  Anti-T antibody, S-: number analyzed (Participants) | 43
  Anti-T antibody, S- | 38
  Anti-T antibody, S+: number analyzed (Participants) | 398
  Anti-T antibody, S+ | 338
  Anti-T antibody, Overall | 376

5. Secondary Outcome: Number of Subjects With a Booster Response to the PT, FHA and PRN Antigens.
Description: Booster response to PT, FHA and PRN antigens was defined according to pre-vaccination antibody concentrations:
  1. for subjects with pre-vaccination values below (<) the assay cut-off, post-vaccination antibody concentration ≥ 4 times the assay cut-off; and
  2. for subjects with pre-vaccination values between the assay cut-off and <4 times the assay cut-off, post-vaccination antibody concentration ≥ 4 times the pre-vaccination antibody concentration; and for subjects with pre-vaccination antibody concentration ≥ 4 times the assay cut-off, post-vaccination antibody concentration ≥ 2 times the pre-vaccination antibody concentration.
  Seronegative (S-) subjects are those who have antibody concentration less than (<) assay cut-off and seropositive (S+) subjects are those who have antibody concentration ≥ assay cut-off prior to vaccination. Assay cut-off was 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti- FHA and 2.187 IU/mL for anti-PRN respectively.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 442
Participants
  Anti-PT antibody, S-: number analyzed (Participants) | 158
  Anti-PT antibody, S- | 138
  Anti-PT antibody, S+ (< 4*assay cut-off): number analyzed (Participants) | 159
  Anti-PT antibody, S+ (< 4*assay cut-off) | 140
  Anti-PT antibody, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 121
  Anti-PT antibody, S+ (≥ 4*assay cut-off) | 97
  Anti-PT antibody, Overall: number analyzed (Participants) | 438
  Anti-PT antibody, Overall | 375
  Anti-FHA antibody, S-: number analyzed (Participants) | 8
  Anti-FHA antibody, S- | 8
  Anti-FHA antibody, S+ (< 4*assay cut-off): number analyzed (Participants) | 57
  Anti-FHA antibody, S+ (< 4*assay cut-off) | 57
  Anti-FHA antibody, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 377
  Anti-FHA antibody, S+ (≥ 4*assay cut-off) | 345
  Anti-FHA antibody, Overall | 410
  Anti-PRN antibody, S-: number analyzed (Participants) | 68
  Anti-PRN antibody, S- | 57
  Anti-PRN antibody, S+ (< 4*assay cut-off): number analyzed (Participants) | 121
  Anti-PRN antibody, S+ (< 4*assay cut-off) | 114
  Anti-PRN antibody, S+ (≥ 4*assay cut-off): number analyzed (Participants) | 245
  Anti-PRN antibody, S+ (≥ 4*assay cut-off) | 225
  Anti-PRN, Overall: number analyzed (Participants) | 434
  Anti-PRN, Overall | 396

6. Secondary Outcome: Anti-D, Anti-T, Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations , One Month After Vaccination.
Description: Antibody concentrations are presented as Geometric Mean Concentrations (GMCs) and expressed in IU/mL. The cut-off for the assays were: 0.057 IU/mL for anti-D, 0.043 IU/mL for anti-T, 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN, respectively.
Time Frame: At Day 31
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | dTpa Group
Number analyzed (Participants) | 442
IU/mL
  Anti-D antibody: number analyzed (Participants) | 438
  Anti-D antibody | 6.287 [5.643 to 7.004]
  Anti-T antibody: number analyzed (Participants) | 441
  Anti-T antibody | 13.507 [12.138 to 15.031]
  Anti-PT antibody: number analyzed (Participants) | 440
  Anti-PT antibody | 59.279 [52.907 to 66.418]
  Anti-FHA antibody | 396.938 [362.876 to 434.197]
  Anti-PRN antibody: number analyzed (Participants) | 436
  Anti-PRN antibody | 249.638 [213.233 to 292.258]

7. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain, redness, swelling. Any = Occurrence of any local symptom regardless of its intensity grade. Any redness and swelling were defined as > 0 millimeters (mm) diameter for all subjects.
Time Frame: During the 4-day (Day 1-4) follow-up period after vaccination.
Population: Analysis was performed on Total Vaccinated Cohort (TVC) which included all subjects with the study vaccine administration and solicited symptoms documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 447
Participants
  Pain | 284
  Redness | 207
  Swelling | 174

8. Secondary Outcome: Number of Subjects Aged Below 6 Years With Solicited General Symptoms.
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness, Loss of appetite and Fever. Any = Occurrence of any general symptom regardless of its intensity grade and relationship to the study vaccination. Fever was defined as temperature ≥ 38.0 degrees Celsius (°C). The location for measuring temperature was the axilla.
Time Frame: During the 4-day (Day 1-4) follow-up period after vaccination.
Population: Analysis was performed on subset of TVC which included subjects aged below 6 years, with the study vaccine administration documented and had solicited symptoms documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 18
Participants
  Drowsiness | 1
  Irritability/Fussiness | 5
  Loss of appetite | 3
  Fever ( ≥ 38°C) | 0

9. Secondary Outcome: Number of Subjects Aged 6 Years and Above With Solicited General Symptoms.
Description: Assessed solicited general symptoms were Fatigue, Gastrointestinal symptoms (included nausea, vomiting, diarrhoea and/or abdominal pain), Headache and Fever. Any = Occurence of any general symptom regardless of its intensity grade and relationship to the study vaccination. Fever was defined as axilla temperature ≥ 38 °C.
Time Frame: During the 4-day (Day 1-4) follow-up period after vaccination.
Population: Analysis was performed on subset of TVC which included subjects aged above and equal to 6 years, with the study vaccine administration documented and had solicited symptoms documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 429
Participants
  Fatigue | 126
  Gastrointestinal symptoms | 34
  Headache | 107
  Fever ( ≥ 38°C), Overall | 10

10. Secondary Outcome: Number of Subjects With Large Swelling Reactions.
Description: Large injection site reaction for subjects < 6 years of age defined as a swelling with a diameter of > 50 mm and for subjects ≥ 6 years of age swelling with a diameter of > 100 mm, noticeable diffuse swelling or noticeable increase in limb circumference. Any = Occurence of any large swelling regardless of its intensity grade and relationship to the study vaccination.
Time Frame: During the 4-day (Day 1-4) follow-up period after vaccination.
Population: Analysis was performed on TVC which included all subjects with the study vaccine administration and solicited symptoms documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 447
Participants | 1

11. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: Any unsolicited AE was defined as any AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Time Frame: During the 31-day (Day 1-31) follow-up period after vaccination
Population: Analysis was performed on TVC which included all subjects with the study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 447
Participants | 52

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 to Day 31
Population: Analysis was performed on TVC which included all subjects with the study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | dTpa Group
Number analyzed (Participants) | 447
Participants | 1

ADVERSE EVENTS:
Time Frame: Unsolicited adverse events (AEs) were reported during the 31-day follow-up period after vaccination. Serious adverse events were reported during the whole study period (from Day 1 up to study conclusion at Day 31).
Description: Solicited adverse events were not reported in this section. They were defined for both age strata (subjects less than 6 years of age and subjects 6 years of age and above), and then, analyzed per age stratum. Please refer to the outcomes section for the results.
Arm/Group | dTpa Group
All-Cause Mortality (participants affected / at risk) | 0/447
Serious Adverse Events (participants affected / at risk) | 1/447
Other Adverse Events (participants affected / at risk) | 52/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=447)
Pneumonia bacterial (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | dTpa Group (N=447)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Induration (General disorders) | 1 (1)
Injection site lymphadenopathy (General disorders) | 1 (1)
Injection site oedema (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 2 (2)
Pyrexia (General disorders) | 3 (3)
Vaccination site erythema (General disorders) | 1 (1)
Vaccination site haematoma (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 7 (7)
Sinusitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 3 (3)
Varicella (Infections and infestations) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (2)
Body temperature increased (Investigations) | 2 (2)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 12 (12)
Somnolence (Nervous system disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT03311659/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/59/NCT03311659/SAP_001.pdf